CLINICAL TRIAL: NCT01152723
Title: Single-dose Pharmacokinetics With Two New Oral Nicotine Replacement Products and Nicorette® Gum. A Study in Healthy Smokers.
Brief Title: Pharmacokinetics With Two New Oral Nicotine Replacement Products and Nicorette® Gum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICTDP1068 (A6431123); 2007-005807-17 (EudraCT Number)
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation, Nicotine pharmacokinetics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- UNG-GA (Experimental): New NRT product
  Interventions: Drug: Nicotine
- UNG-GB (Experimental): New NRT product
  Interventions: Drug: Nicotine
- Nicorette® Gum (Active Comparator): Nicorette® Gum
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — 2 mg, Single Dose
  Other Names: Experimental NRT UNG-GA and UNG-GB, and Nicorette® Gum

SUMMARY:
Single-dose pharmacokinetics with two new oral nicotine replacement products and Nicorette® gum.

DETAILED DESCRIPTION:
The study is a single-dose, randomized, cross-over study. The investigational products will be given as single doses at separate visits. The product administrations comprise 30 minutes of chewing. Periods without NRT, lasting for at least 36 hours, will separate treatment visits. Before and after the start of product administration at each treatment visit, blood will be sampled for pharmacokinetic analyses, pre-dose, and during 8 hours after start of product administration. Used gums will be collected and analyzed to determine the amount of remaining nicotine. Subjects will also be monitored to capture any adverse events that may occur. Treatment labels will be concealed from subjects and study personnel.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, smoking at least 10 cigarettes daily during at least one year preceding inclusion and BMI between 17.5 and 30.0 kg/m2.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product or donation or loss of blood within 3 month preceding the first dose of study medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic measurements | Baseline and during 8 hours after product administration
  Pharmacokinetic measurements including:
  * the maximum observed nicotine concentration in plasma (Cmax)
  * the area under the plasma concentration-vs.-time curve until the last measurable concentration (AUCt)
  * the area under the plasma concentration-vs.-time curve until infinity (AUC∞)

SECONDARY OUTCOMES:
tmax | During 8 hours after start of product administration
  The time of occurrence of Cmax following product administration
Lamda z | During 8 hours after start of product administration
  The terminal nicotine elimination rate constant (λz)
Released amount of nicotine | After 30 minutes of chewing
  The amount of nicotine released from gums during 30 minutes' chewing.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- McNeil AB Clinical Pharmacology R&D, Lund, Sweden